CLINICAL TRIAL: NCT05659797
Title: Pilot Study Evaluating the Uptake of [18F]Fluoroestradiol (FES) BPET/DBT in Primary Breast Cancer to Measure the Localized Extent of Estrogen Receptor Positive Disease
Brief Title: FES BPET-DBT in Newly Diagnosed Breast Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UPCC 08122; 852000 (Other: Abramson Cancer center)
Record Dates: First submitted 2022-12-05; First posted 2022-12-21 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: PET; 18F-Fluoroestradiol
MeSH Terms: conditions — Breast Neoplasms | interventions — 16-fluoroestradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- FES BPET-DBT (Experimental): FES-BPET/DBT imaging session
  Interventions: Device: BPET/DBT imaging; Drug: 18F-FES

INTERVENTIONS:
Device: BPET/DBT imaging — Imaging of the breast with a novel device combining dedicated Breast Positron Emission Tomography (BPET) and Digital Breast Tomosynthesis (DBT) following intravenous injection of [18F]-Fluoroestradiol (FES).
Drug: 18F-FES — Radiolabelled fluoroestradiol for PET imaging
  Other Names: 18F-fluoroestradiol

SUMMARY:
Patients with newly diagnosed primary estrogen-receptor (ER) positive breast cancer, with at least one breast lesion that is 1.0 cm in diameter or greater, may be eligible for this study. Patients may participate in this study if they are at least 18 years of age. Up to 20 evaluable subjects will participate in a single imaging cohort. Study subjects will undergo imaging of the breast with a novel device combining dedicated Breast Positron Emission Tomography (BPET) and Digital Breast Tomosynthesis (DBT) following intravenous injection of [18F]-Fluoroestradiol (FES). This is an observational study; FES-BPET/DBT will not be used to direct treatment decisions. While patients and referring physicians will not be blinded to the FES-BPET/DBT results, treatment decisions are made by the treating physicians based upon standard clinical imaging.

DETAILED DESCRIPTION:
The FES-BPET/DBT imaging session will include an injection of approximately 6 mCi (expected range of injected dose is 3-7 mCi) FES. Pilot data will be collected to evaluate image quality of FES-BPET/DBT in primary breast cancer. Size and focality of breast cancer extent as measured by FES-BPET/DBT will be compared to disease extent on standard breast imaging modalities. FES uptake on BPET/DBT, as measured by SUV, will be compared to ER expression by immunohistochemistry (IHC) on biopsy specimens. In addition, all subjects in this study will be recruited to the open ended Penn protocol titled 'Evaluation of Long-Axial Field-of-View Positron Emission Tomography Scanner,' IRB #843546. In those subjects who consent to this proposed study as well as #843546, assessment of disease extent on FES-BPET/DBT will be compared to that on whole body PET. Of note, those subjects who also consent to #843546 will not undergo any additional injected dose of FES radiotracer. This preliminary study seeks to evaluate FES-BPET/DBT as a preoperative imaging assay of ER-positive breast cancer disease extent within the breast.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be ≥ 18 years of age.
2. Known ER positive (by immunohistochemistry) breast cancer.
3. At least one lesion ≥ 1.0 cm that is seen on standard imaging (e.g. mammogram, ultrasound, MRI, CT, FDG-PET/CT). Only one type of imaging is required to show a lesion.
4. Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

1. Females who are pregnant or breast feeding will not be eligible for this study; a urine pregnancy test will be performed in women of child-bearing potential prior to PET imaging..
2. Inability to tolerate imaging procedures in the opinion of an investigator or treating physician.
3. Currently taking tamoxifen or raloxifene
4. Any current medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician investigator to be a condition that could compromise participant safety or successful participation in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Uptake of FES on BPET | 6 weeks
  Different types of SUV measurements (e.g. Max, Mean and Peak) may be tested to identify the optimal method for analyses for future studies of FES-BPET/DBT.
Image quality | 6 weeks
  The image quality of the study DBT will be compared to the clinical DBT in terms of image quality
Image artifacts | 6 weeks
  Image artifacts on study DBT will be compared to clinical DBT
Parenchymal appearance | 6 weeks
  The parenchymal appearance of the study DBT will be compared to the clinical DBT
Tumor size and extent | 6 weeks
  The size/extent of tumor on the study DBT will be compared to the clinical DBT

SECONDARY OUTCOMES:
Estrogen receptor IHC | 8 weeks
  Clinical immunohistochemical estrogen receptor (ER) results from biopsy or surgery will be compared to FES PET uptake

CONTACTS AND LOCATIONS:
Overall Officials: Christine Edmonds, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States